CLINICAL TRIAL: NCT03502265
Title: Exploring Otteroo Use In Early Intervention: A Case Series
Brief Title: Otteroo Case Series
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Beth A. Smith, Assistant Professor, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-17-00910
Record Dates: First submitted 2018-04-03; First posted 2018-04-18 (Actual); Results first posted 2021-10-27 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-10

CONDITIONS: Infants With or at Risk/Concern for Developmental Delay

STUDY DESIGN:
Intervention Model Description: single subject research design case series
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Otteroo adjunct (Experimental): A single-subject research design will be used: measures of infant development will be collected across a 4-week baseline period (standard care), 4 weeks of intervention (standard care and Otteroo use), and a 4 weeks of reversal/retention period (standard care). There is only one arm due to the study design. It is a within-subjects comparison, not a between-subjects comparison of different study arms.
  Interventions: Other: Otteroo

INTERVENTIONS:
Other: Otteroo — Otteroo will be provided for 4 weeks of use, to supplement any standard care. Standard care is not provided.

SUMMARY:
Rationale. The Otteroo is a floatie which supports an infant or young child with their head above and their body in water. Researchers are proposing that the Otteroo may be a good "tool" to facilitate exploring the ability to move and control one's body before locomotion develops. Intervention. Otteroo will be used as an adjunct to standard care for 4 weeks.

DETAILED DESCRIPTION:
Objectives or purpose. The purpose of this project is to measure overall developmental status before, during, and after Otteroo experience. Study population or sample characteristics. Participants will be 4 pre-locomotor infants or young children for whom a healthcare provider or caregiver has identified concerns about potential developmental delay. Study methodology. A single-subject research design will be used: measures of infant development will be collected across a 4-week baseline period (standard care), 4 weeks of intervention (standard care and Otteroo use), and a 4 weeks of reversal/retention period (standard care). Study endpoints or outcomes. The end of the study is the final assessment at 12 weeks. Follow-up. None. Statistics and plans for analysis. Researchers will calculate descriptive statistics (mean, range, coefficient of variation) for all measures and describe changes over time, relating the participant's performance at each time point to norm-referenced results for their age.

ELIGIBILITY:
Inclusion Criteria:

* pre-locomotor (able to locomote independently less than 4 feet)
* a healthcare provider or caregiver has identified concerns about potential developmental delay

Exclusion Criteria:

* younger than 8 weeks of age
* older than 66 months of age
* body weight of more than 35 lbs
* diagnosis of Down syndrome
* clinical presentation of ligamentous laxity
* without access to an appropriate water source (bathtub or pool depending on the size of the child)
* with prior experience using Otteroo

Ages: 8 Weeks to 66 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Infant Neuromotor Control Laboratory, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
available upon request from the PI (Beth Smith)
Supporting Information: Study Protocol, SAP, ICF
Time Frame: available for 3 years following publication of results in peer-reviewed journal
Access Criteria: available upon request from the PI (Beth Smith) at beth.smith@usc.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Otteroo Adjunct
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Otteroo Adjunct
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: days] | 403 (353)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4
Alberta Infant Motor Scale [Mean (Full Range); unit: overall percentile score (range 0-100)] — Observational scale of motor skills. Full percentile range is 0-100%. A score of 30% means a child is ahead of 30% of children the same age and behind 70% of children the same age. A score of 80% means a child is ahead of 80% of children the same age and behind 20% of children the same age.
  overall percentile score (range 0-100) | 11 [5 to 25]

OUTCOME MEASURES:

1. Primary Outcome: Change in Alberta Infant Motor Scale
Description: observational scale of motor skills, change in percentile score from week 0 to week 12 for each child. Full percentile range is 0-100%. Change of 0 means no change in percentile score, change of 100 means child went from 0% to 100% or 100% to 0% which is the maximum possible change in percentile score. A positive change means the percentile increased, while a negative change means the percentile decreased.
Time Frame: weeks 0 and 12
Measure: Mean (Full Range); unit: change in percentile
Arm/Group | Otteroo Adjunct
Number analyzed (Participants) | 4
change in percentile | 5 [-5 to 25]

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Otteroo Adjunct
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-08): https://cdn.clinicaltrials.gov/large-docs/65/NCT03502265/Prot_SAP_000.pdf